CLINICAL TRIAL: NCT07149662
Title: B-cellspåverkan i Barn Till Kvinnor Med Multipel Skleros Och Rituximabbehandling före Eller Under Graviditeten (B-cell Effects in Children Born to Women With Multiple Sclerosis and Rituximab Treatment Before or During Pregnancy)
Brief Title: Immune System Effects in Children Born to Women With Multiple Sclerosis Treated With Monoclonal Antibody Therapy During Pregnancy
Status: Not yet recruiting | Type: Observational
Sponsor: Region Stockholm (Other Government)
Collaborators: The Swedish Research Council (Other Government); Haukeland University Hospital (Other); Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Katharina Fink, MD, Dr. med., Region Stockholm
Other Study IDs: 2024-00763-02
Record Dates: First submitted 2025-07-30; First posted 2025-09-02 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-08

CONDITIONS: Multiple Sclerosis; Pregnancy
Keywords: Multiple Sclerosis; Rituximab; Ocrelizumab; Ofatumumab; monoclonal CD-20 antibodies; Pregnancy
MeSH Terms: conditions — Multiple Sclerosis | interventions — Rituximab; ocrelizumab; ofatumumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Women with MS during pregnancy: Women over 18 years of age with the diagnosis of multiple sclerosis, regardless of treatment, or no treatment, that have successfully delivered or will deliver a child
  Interventions: Drug: monoclonal CD-20 antibodies; Drug: No Drug; Drug: Other treatment
- Infants born to women with MS: Infants born to women with multiple sclerosis
  Interventions: Drug: monoclonal CD-20 antibodies; Drug: No Drug; Drug: Other treatment

INTERVENTIONS:
Drug: monoclonal CD-20 antibodies — Treatment with monoclonal CD-20 antibodies 6 months before or during pregnancy
  Other Names: rituximab; ocrelizumab; ofatumumab
Drug: No Drug — No medication
Drug: Other treatment — Any other immune modulating treatment

SUMMARY:
The goal of this observational study is to learn about consequences for the child when the mother is treated with rituximab (or other monoclonal CD-20 antibodies) before or during pregnancy. The main questions it aims to answer are:

* Is the infant's immune system effected with lower levels of B-cell markers, higher rates of infections or poor vaccine response?
* Are the monoclonal CD20-antibodies fully eliminated in women treated within 6 (12) months prior to conception?

Participants will:

* At the time of clinical routine blood sampling (at the end of each trimester) the becoming mother will give some additional blood samples for analysis of drug concentration
* Within the first year postpartum the child will leave a blood sample to detect antibodies induced by vaccination or infections
* Within our routine contacts with the participant (mother) will be asked about infections in both the mother and the child

DETAILED DESCRIPTION:
In offspring to women with MS and current pregnancies the investigators will address if a reduction in the levels of KREC (kappa-deleting recombination excision circles) and/or CD19+ B-cells at birth has clinical significance. Participants with MS regardless of treatment that have successfully delivered or will deliver a child will be asked for informed consent and after given informed consent they will be included in the study.

1. At the time of clinical routine sampling in the becoming mother the investigators will collect additional blood samples. Routine analysis collects information on immunoglobulin levels and b-cell levels, additional blood samples will allow analysis of drug concentration at the end of every trimester.
2. Within the first year postpartum, but earliest one month after vaccination, the investigators will ask for a blood sample from the child to detect antibodies induced by vaccination or infections to secure the ability to develop antibodies despite being exposed to monoclonal CD20-antibodies in-utero or via breastmilk. All children followed by the Specialist outpatient clinic for children in Liljeholmen - a specialist clinic from the Karolinska University Hospital following children to mothers on immunosuppressant/immunomodulating treatments regardless of disease, will be offered blood sampling by routine months 2, 6 and 1 year postpartum. In collaboration with this center, the investigators will get samples taken and analyzed within clinical routine.
3. PKU-test is taken in the child within routine but additional analysis on drug levels and KREC will be analyzed as well as determining abundance of CD19 transcripts.
4. Within the routine contacts with the MS patient (mother) the investigators will ask for infections in both, the mother and the child at 3 months and 1 year post-partum.

ELIGIBILITY:
Inclusion Criteria:

* Established multiple sclerosis diagnosis
* Rituximab, ocrelizumab, ofatumumab or other monoclonal CD-20 antibody has been administered within 6 (12) months prior to or during pregnancy
* Other immun modulation treatment has been administered within 6 (12) months prior to or during pregnancy
* No treatment has been administered within 6 (12) months prior to or during pregnancy

Exclusion Criteria:

- Previous stem cell transplantation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Able to become pregnant and deliver a child
Study Population: Women diagnosed with multiple sclerosis that are patients at the Academic specialist center, Center for Neurology, Stockholm, Sweden
Sampling Method: Non-Probability Sample
Enrollment: 111 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-10 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Effect on infant immune system | At birth
  Levels of KREC (copies/micro L) at birth.
Effect on infant immune system | At birth
  CD19+ B-cell (nx10^9 cells/L) levels at birth
Effect on infant immune system | Age 2 months - 1 year
  Infant levels of antibodies (g/L) induced by vaccination or infections
Effect on infant immune system | Age 1 year
  Infection during first year of life (n/12 months)

SECONDARY OUTCOMES:
Drug level concentration infant | At birth - 3 days old
  Drug level concentration (microgram/ml) measured from dried blood spots (PKU-test)

OTHER OUTCOMES:
Effects on mother´s immune system | From enrollment to three months after birth
  Immunoglobulin (g/L) levels
Effects on mother´s immune system | From enrollment to three months after birth
  B-cell levels nx10^9/L
Effects on mother´s immune system | From enrollment to three months after birth
  Drug concentration (microgram/ml)

CONTACTS AND LOCATIONS:
Overall Officials: Katharina Fink, MD, Dr. med., Study Director — Karolinska Institutet
Locations (1):
- Academic specialist center, Center for Neurology, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Yes
We plan to share all pseudoanonymised IPD that underlie results in a future publication.